CLINICAL TRIAL: NCT01190319
Title: Effect of Strawberry Powder on Blood Pressure in Individuals With Pre-Hypertension
Brief Title: Study: Effects of Strawberries on Blood Pressure
Acronym: CSCBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: California Strawberry Commission (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 200715153
Record Dates: First submitted 2009-10-20; First posted 2010-08-27 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Pre-hypertension
Keywords: blood pressure; strawberry; fruit phenolics; LDL oxidation; Flow mediated dilation (FMD)
MeSH Terms: conditions — Prehypertension | interventions — Beverages

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo Beverage (Placebo Comparator): The placebo beverage is matched in energy, macronutrient composition and sensory properties to the active beverage, but is devoid of strawberry polyphenols.
  Interventions: Other: Placebo
- Strawberry Beverage (Experimental): The strawberry beverage is matched in energy, macronutrient composition and sensory properties to the placebo beverage, but contains strawberry polyphenols.
  Interventions: Other: Strawberry Beverage

INTERVENTIONS:
Other: Strawberry Beverage — Beverage, daily for 8 weeks, 12g freeze-dried strawberry powder
  Other Names: Strawberry powder made from a mix of California strawberries.
  Arms: Strawberry Beverage
Other: Placebo — Placebo beverage, 8 weeks
  Other Names: Beverage
  Arms: Placebo Beverage

SUMMARY:
The specific aim of the study is to determine whether a freeze dried powder provided by the California Strawberries Commission, can reduce blood pressure in patients with pre-hypertension. The powder is prepared by the California Strawberry Commission (CSC).

DETAILED DESCRIPTION:
Primarily, we would like to find out whether freeze dried strawberry powder lowers blood pressure. In addition we would like to know if the strawberry alters the subject's blood cholesterol and the ability of the subject's blood vessels to relax.

ELIGIBILITY:
Inclusion Criteria:

* Pre-hypertensive men and women (JNC 7 [The Seventh Report of the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure] criteria) between the ages of 25 and 65 years who have no clinical evidence/history of cardiovascular, respiratory, renal, gastrointestinal or hepatic disease.

Exclusion Criteria:

* Subjects who:

  1. are taking over the counter anti-oxidant supplements,
  2. are taking prescription medications that may interfere with study procedures or endpoints,
  3. have unusual dietary habits (eg., pica),
  4. are actively losing weight or trying to lose weight,
  5. are addicted to drugs or alcohol,
  6. present with significant psychiatric or neurological disturbances,
  7. have known allergies to strawberry, will be excluded from participating in this study.
  8. Patients known to have glaucoma
  9. Pregnant and/or lactating females

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-09 (Actual); Primary Completion 2011-10 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in blood pressure | 8 weeks

SECONDARY OUTCOMES:
Change in low density lipoprotein (LDL) oxidation | 8 weeks
Change in flow mediated dilation (FMD) | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Chulani T Kappagoda, MD, Principal Investigator — University of California, Davis; Britt Burton-Freeman, Ph.D, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis (Ragle Hall), Davis, California, United States